CLINICAL TRIAL: NCT00378742
Title: National Ophthalmic Genotyping and Phenotyping Network Stage 1 - Creation of DNA Repository for Inherited Ophthalmic Diseases
Brief Title: Repository for Inherited Eye Diseases
Status: Completed | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060236; 06-EI-0236
Record Dates: First submitted 2006-09-20; First posted 2006-09-21 (Estimated); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Retinitis Pigmentosa; Inherited Ophthalmic Diseases
Keywords: Macular Dystrophy; Phenotype-Genotype correlation; Genetics; Retinitis Pigmentosa; Inherited; Natural History
MeSH Terms: conditions — Retinitis Pigmentosa; Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: Participants with inherited eye diseases or relative of affected participant

SUMMARY:
The National Ophthalmic Disease Genotyping and Phenotyping Network (eyeGENE(R)) is a genomic medicine initiative created by the National Eye Institute (NEI), part of the National Institutes of Health (NIH), in partnership with clinics and laboratories across the vision research community. The core mission of eyeGENE(R) is to facilitate research into the causes and mechanisms of rare inherited eye diseases and accelerate pathways to treatments. This study collects DNA samples from patients with inherited eye diseases to facilitate research to identify genetic factors responsible for these conditions. Nearly 500 genes that contribute to inherited eye diseases have been identified. As a result, gene-based therapies are being pursued to treat eye genetic diseases that were once considered untreatable.

Physicians in collaborating institutions will recruit patients to participate in the study. Patients will provide a blood sample and undergo a standard eye examination. The blood sample and clinical information will then be sent to the NEI for testing, processing and storing in the biorepository. Patients are given the option to receive results back and/or to be re-contacted in the event of future clinical studies. Information supplied to the testing laboratories includes a unique identification number, the patient gender, and the patient date of birth. The stored samples are available to researchers along with information about the patient's disease, but without patient identifiers.

DETAILED DESCRIPTION:
Molecular genetics has the potential to revolutionize the diagnosis and treatment of inherited eye diseases. Progress in research on inherited eye disease would be augmented by the availability of patient DNA coupled to robust, anonymous phenotypic information. The National Ophthalmic Genotyping and Phenotyping Network (eyeGENE(R)) has been created to answer this need. By creating a national DNA and blood repository for inherited eye disease. These samples have been gathered from clinical centers around the nation and will be coupled to anonymous, phenotypic descriptors. If requested, a portion of the sample submitted by a clinician can be used for appropriate, CLIA-certified molecular diagnostics that can be used in patient care. Once a sufficient repository is created, researchers will be able to request aliquots for their laboratory experiments. Participants will be provided the option to be re-contacted if an approved clinical study for which they might qualify is offered. Researchers can request aliquots for their laboratory experiments or ask the eyeGENE(R) Coordinating Center to re-contact participants to inform them about the possibility to participate in a clinical study.

ELIGIBILITY:
* INCLUSION CRITERIA:

To participate in this protocol:

1a. The participant must present with characteristics that meet minimal clinical criteria established by eyeGENE, as determined by the referring clinician.

OR

1b. The participant must be a relative of an affected participant if analysis would help with the interpretation of an affected participant's test results or to obtain some useful information as decided by the eyeGENE Research Study Group.

2. The participant must be willing and able to provide a suitable blood sample.

EXCLUSION CRITERIA:

* Severe systemic disease that compromise the ability of the referring clinician to obtain an adequate eye examination.
* Any disease or condition that makes it unsafe for a subject to provide a blood sample of at least 5 ml for children and at least 15ml for adults.
* Inability to cooperate with phlebotomy and clinical examination.
* Those with impaired decision-making capability who do not have a legally-authorized representative.
* If clinical criteria information, consent forms, or a blood sample can not be provided by the doctor or participant after one year of submitting a blood sample to eyeGENE .

Ages: 1 Day to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with inherited eye diseases or their unaffected relatives.
Sampling Method: Non-Probability Sample
Enrollment: 6618 (Actual)
Dates: Start 2006-09-20 (Actual); Primary Completion 2015-11-19 (Actual); Study Completion 2015-11-19 (Actual)

PRIMARY OUTCOMES:
Obtain samples for the creation of eyeGENE network | 34 years
  Obtain and create a national DNA and blood repository for inherited eye diseases.

CONTACTS AND LOCATIONS:
Overall Officials: Brian P Brooks, M.D., Principal Investigator — National Eye Institute (NEI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bender C, Woo EG, Guan B, Ullah E, Feng E, Turriff A, Tumminia SJ, Sieving PA, Cukras CA, Hufnagel RB. Predominant Founder Effect among Recurrent Pathogenic Variants for an X-Linked Disorder. Genes (Basel). 2022 Apr 12;13(4):675. doi: 10.3390/genes13040675. PMID 35456481
- [Derived] Parrish RS, Garafalo AV, Ndifor V, Goetz KE, Reeves MJ, Yim A, Cooper RC, Iano-Fletcher J, Wang X, Tumminia SJ. Sample Confirmation Testing: A Short Tandem Repeat-Based Quality Assurance and Quality Control Procedure for the eyeGENE Biorepository. Biopreserv Biobank. 2016 Apr;14(2):149-55. doi: 10.1089/bio.2015.0098. Epub 2016 Feb 18. PMID 26891080
- [Derived] Alapati A, Goetz K, Suk J, Navani M, Al-Tarouti A, Jayasundera T, Tumminia SJ, Lee P, Ayyagari R. Molecular diagnostic testing by eyeGENE: analysis of patients with hereditary retinal dystrophy phenotypes involving central vision loss. Invest Ophthalmol Vis Sci. 2014 Jul 31;55(9):5510-21. doi: 10.1167/iovs.14-14359. PMID 25082885
- [Derived] Sullivan LS, Bowne SJ, Reeves MJ, Blain D, Goetz K, Ndifor V, Vitez S, Wang X, Tumminia SJ, Daiger SP. Prevalence of mutations in eyeGENE probands with a diagnosis of autosomal dominant retinitis pigmentosa. Invest Ophthalmol Vis Sci. 2013 Sep 19;54(9):6255-61. doi: 10.1167/iovs.13-12605. PMID 23950152
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2006-EI-0236.html